CLINICAL TRIAL: NCT00406718
Title: Interventions for Adherence to Oral Antipsychotic Medications in Schizophrenia
Brief Title: Improving Adherence to Oral Antipsychotic Medications in People With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Dawn Velligan, Clinical Professor Department of Psychiatry, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH074047 (NIH)
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Results first posted 2015-10-05 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-07

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Medication Adherence; Psychosocial Treatment; Cognitive Adaptation Training; Med-e Monitor; Adaptive Function
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Medication Adherence | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- PharmCAT (Experimental): Participants will receive PharmCAT in addition to Treatment as usual, Pharm CAT is a psychosocial intervention using environmental supports such as signs, alarms, checklists, and special medication containers to cue and sequence adaptive behavior in the patient's home environment. This treatment specifically targets adherence to medication, medication education, and orientation for patients with schizophrenia. Participants will receive weekly home visits from a case manager.
  Interventions: Behavioral: PharmCAT
- Med-eMonitor (Active Comparator): Participants will receive Med-eMonitor™ in addition to treatment as usual. Participants will use the Med-eMonitor™ device, which is an electronic device that holds up to one month's supply of up to five medications. It is capable of cueing the taking of medication, warning patients when they are taking the wrong medication or taking it at the wrong time, recording side effect complaints, and through modem hookup promptly alerting treatment staff of failures to take medication as prescribed.
  Interventions: Behavioral: Med-eMonitor
- Treatment as Usual (Active Comparator): Participants will receive standard treatment as usual which is medication management and limited case management provided by the CMHC.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Med-eMonitor — Participants will use the Med-eMonitor™ device, which is an electronic device that holds up to one month's supply of up to five medications. It is capable of cueing the taking of medication, warning patients when they are taking the wrong medication or taking it at the wrong time, recording side effect complaints, and through modem hookup promptly alerting treatment staff of failures to take medication as prescribed.
  Arms: Med-eMonitor
Behavioral: PharmCAT — Pharm CAT is a psychosocial intervention using environmental supports such as signs, alarms, checklists, and special medication containers to cue and sequence adaptive behavior in the patient's home environment. This treatment specifically targets adherence to medication, medication education, and orientation for patients with schizophrenia. Participants will receive weekly home visits from a case manager.
  Arms: PharmCAT
Behavioral: Treatment as Usual — Participants receiving standard treatment will keep the Med-eMonitor™ device in their homes throughout the study but will not use its medication reminder function.
  Arms: Treatment as Usual

SUMMARY:
This study will determine the comparative effectiveness of two systems designed to improve medication adherence in people with schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is a severely debilitating mental disorder. People with schizophrenia often experience unusual thoughts or perceptions, decreased pleasure in everyday life, and difficulty functioning in social situations. Antipsychotic medications have been shown to be effective in improving the symptoms of schizophrenia. Poor adherence to medication, however, leads to re-hospitalization, impedes the process of recovery, and contributes to the high costs associated with schizophrenia treatment. Studies have shown that PharmCAT, cognitive adaptive training that specifically targets medication adherence, has been effective in improving adherence and outcomes in people with schizophrenia. The Med-eMonitor™ is a new pill device that is able to alert patients when they should take medication, when they are taking the wrong medication, and when they are taking medication at the wrong time. The device can also record side effect complaints and then send stored information to treatment staff. The capabilities of the Med-eMonitor™ eliminate the need for the weekly home visits that are necessary in the PharmCAT program, and may make treatment more easily available to individuals in remote or rural settings. This study will compare the effectiveness of PharmCAT, the Med-eMonitor™, and standard treatment in improving medication adherence and treatment outcome in people with schizophrenia.

Participants in this study will be randomly assigned to one of the following treatment groups: (1) PharmCAT; (2) the Med-eMonitor™; or (3) standard treatment. Participants in Group 1 will receive weekly home visits from a case manager. These visits will specifically target medication adherence. Participants in Group 2 will use the Med-eMonitor™ device. Data recorded by the device will be sent electronically to study staff. Participants in Group 3 will keep the Med-eMonitor™ device in their homes throughout the study but will not use its medication reminder function. The device will record only when medication is taken. All participants will report to the study site at study entry and Months 4, 7, and 10 for measures of symptoms, functioning, social activities, and relationships.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder according to DSM-IV criteria, as determined on the basis of the Structured Clinical Interview for Diagnosis (SCID-P)
* Receiving treatment with an oral atypical antipsychotic medication other than clozapine (e.g., risperidone, olanzapine, quetiapine, aripiprazole, ziprasidone, or others as they are FDA approved)
* Assumes some responsibility for taking own medications
* Able to provide evidence of a stable living environment (e.g., individual apartment, family home, or board and care facility) within 3 months prior to study entry and no plans to move in the next year
* Intact visual and auditory ability as determined by a computerized screening battery
* Ability to read at the 5th grade level or higher based upon score on the Wide Range Achievement Test (WRAT)
* Able to understand and complete rating scales and neuropsychological testing
* Working telephone present in the home

Exclusion Criteria:

* History of significant head trauma, seizure disorder, or mental retardation
* Alcohol or drug abuse or dependence within 3 months prior to study entry
* Currently being treated by an assertive community treatment (ACT) team
* History of violence within 1 year prior to study entry
* Any hospitalizations within 3 months prior to study entry

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 197 (Actual)
Dates: Start 2006-11; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn I. Velligan, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio (UTHSCSA)
Locations (1):
- The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 197 signed consents, but only 142 were randomized. 24 no longer wanted to participate, 15 were lost to follow up and could not be contacted, 11 did not meet inclusion criteria once documentation was reviewed, 2 moved out of the area and 3 individuals had family who did not want the individual to participate, leading them to withdraw consent.
Groups:
- Pharm CAT: Pharm CAT is a psychosocial intervention using environmental supports such as signs, alarms, checklists, and special medication containers to cue and sequence adaptive behavior in the patient's home environment. This treatment specifically targets adherence to medication, medication education, and orientation for patients with schizophrenia. Participants will receive weekly home visits from a case manager.
- Med-eMonitor: Participants will receive the Med-eMonitor™
  Med-eMonitor Device: Participants will use the Med-eMonitor™ device, which is an electronic device that holds up to one month's supply of up to five medications. It is capable of cueing the taking of medication, warning patients when they are taking the wrong medication or taking it at the wrong time, recording side effect complaints, and through modem hookup promptly alerting treatment staff of failures to take medication as prescribed.
- Treatment as Usual: standard treatment
  Standard treatment: Participants receiving standard treatment will keep the Med-eMonitor™ device in their homes throughout the study but will not use its medication reminder function.
Period: Overall Study
Arm/Group | Pharm CAT | Med-eMonitor | Treatment as Usual
Started | 47 | 48 | 47
Completed | 43 | 34 | 39
Not Completed | 4 | 14 | 8
Not completed — Withdrawal by Subject | 2 | 9 | 4
Not completed — Lost to Follow-up | 2 | 5 | 4

BASELINE CHARACTERISTICS:
Population: X2 for categorical, and one way anova for continuous to examine differences in demographics for participants not making it to randomization versus those randomized to treatment.
Groups:
- PharmCAT: Participants will receive PharmCAT
  PharmCAT Therapy: Pharm CAT is a psychosocial intervention using environmental supports such as signs, alarms, checklists, and special medication containers to cue and sequence adaptive behavior in the patient's home environment. This treatment specifically targets adherence to medication, medication education, and orientation for patients with schizophrenia. Participants will receive weekly home visits from a case manager.
- Standard Treatment: Participants will receive standard treatment
  Standard treatment: Participants receiving standard treatment will keep the Med-eMonitor™ device in their homes throughout the study but will not use its medication reminder function.
- Total: Total of all reporting groups
Arm/Group | PharmCAT | Med-eMonitor | Standard Treatment | Total
Number analyzed (Participants) | 47 | 48 | 47 | 142
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 47 | 48 | 47 | 142
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.0 (11.04) | 43.0 (10.15) | 42.0 (9.27) | 42.52 (10.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 23 | 68
  Male | 24 | 26 | 24 | 74
Region of Enrollment [Number; unit: participants]
  United States | 47 | 48 | 47 | 142

OUTCOME MEASURES:

1. Primary Outcome: Adherence
Description: Adherence derived from electronic monitoring. Percentage of medication taken during each preceding 3 month period, averaged across treatment period.
Time Frame: Measured at Months 4, 7, and 10 months averaged across the treatment period which began 1 month after study baseline and ended at month 10 (total 9 mos of treatment)
Population: All individuals randomized who had a baseline and at least one follow-up rating
Measure: Mean (Standard Deviation); unit: Percentage of medication taken
Groups:
- Standard: Participants will receive standard treatment
  Standard treatment: Participants receiving standard treatment will keep the Med-eMonitor™ device in their homes throughout the study but will not use its medication reminder function.
Arm/Group | PharmCAT | Med-eMonitor | Standard
Number analyzed (Participants) | 46 | 46 | 45
Percentage of medication taken | 91.84 (11.07) | 88.61 (16.07) | 72.55 (26.84)

2. Primary Outcome: Social and Occupational Functioning Assessment Scale (SOFAS) Scores
Description: Scale from 1-100 rating global social and occupational functioning. Higher scores indicate better functional outcomes
Time Frame: as for outcome 1
Population: Patients with baseline and at least one follow up rating
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PharmCAT | Med-eMonitor | Standard
Number analyzed (Participants) | 46 | 46 | 45
Units on a scale | 91.84 (11.70) | 88.61 (16.07) | 73.19 (25.66)

3. Secondary Outcome: Schizophrenia Symptoms
Description: Brief Psychiatric Rating Scale (BPRS) expanded version psychosis subscale, mean of items for unusual thought content, auspiciousness, conceptual disorganization, and hallucinations. Higher scores mean greater level of symptomatology. Scores vary from 1 = absent to 7 = severe
Time Frame: as for outcome 1
Population: All subjects with a baseline and at least one follow up rating
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pharm CAT | Med-eMonitor | Treatment as Usual
Number analyzed (Participants) | 46 | 46 | 45
units on a scale | 2.73 (.13) | 2.75 (.13) | 2.72 (.13)

ADVERSE EVENTS:
Time Frame: Reported annually in IRB report patients followed only for the 10 month duration of the study.
Arm/Group | PharmCAT | Med-eMonitor | Standard Treatment
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/48 | 0/47
Other Adverse Events (participants affected / at risk) | 0/47 | 1/48 | 0/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PharmCAT (N=47) | Med-eMonitor (N=48) | Standard Treatment (N=47)
paranoia from monitor (Psychiatric disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Patients had long-standing illness and results may not apply to patients with a more recent onset of schizophrenia/schizoaffective disorder

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No